CLINICAL TRIAL: NCT02486393
Title: Complications in Parotid Surgery - a Prospective Cohort Study
Brief Title: Complications in Parotid Surgery
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Leif Bäck, MD PhD, Helsinki University Central Hospital
Other Study IDs: JR/Helsinki/ORL/
Record Dates: First submitted 2015-06-25; First posted 2015-07-01 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Facial Palsy
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- type of surgery: patients undergoing parotid surgery
  Interventions: Procedure: Parotid surgery

INTERVENTIONS:
Procedure: Parotid surgery — Surgery of the parotid gland tumours

SUMMARY:
The investigators conducted a prospective study of 132 patients undergoing benign parotid surgery at our department. Their primary objective was to analyze the incidence of and contributing factors associated with temporary and permanent postoperative facial palsy with strictly standardized methods in facial nerve function evaluation. Also other complications occurring within 12 months of operation were recorded.

DETAILED DESCRIPTION:
Patients who underwent parotid surgery at the Department of Otorhinolaryngology - Head and Neck Surgery, Helsinki University Hospital, Helsinki, Finland, between September 2011 and November 2012 were prospectively enrolled. Exclusion criteria were age under 18, suspicion of malignancy or facial schwannoma, a tumor extending into the parapharyngeal space, and previous parotid surgery exposing facial nerve.

ELIGIBILITY:
Inclusion Criteria:

* parotid gland tumour surgery

Exclusion Criteria:

* age under 18
* suspicion of malignancy or facial schwannoma
* a tumor extending into the parapharyngeal space
* previous parotid surgery exposing facial nerve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent parotid surgery at the Department of Otorhinolaryngology - Head and Neck Surgery, Helsinki University Hospital, Helsinki, Finland, between September 2011 and November 2012 were prospectively enrolled
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
facial palsy | post op 12 months